CLINICAL TRIAL: NCT04676542
Title: The Effects of Externally Paced Exercise on Cognitive Performance and Stress in College Aged Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-1535
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Performance
Keywords: Martial Arts, Walking, Cognitive Performance,Stress
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The proposed research design will be utilizing a randomized cross over repeated measures design. Subjects will take part in two separate conditions: 1) One hour of a beginning martial art class (EP), and 2) One hour walk at 4.0 mph pace (IP).The independent variables are the two conditions and the dependent variables are processing speed, attention, executive function (Stroop Color and Word tests), and a stress visual analog scale
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One group taking part in 2 separate conditions (Experimental): The proposed research design will be utilizing a randomized cross over repeated measures design. Subjects will take part in two separate conditions: 1) One hour of a beginning martial art class (EP), and 2) One hour walk at 4.0 mph pace (IP).
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — One hour of a beginning martial art class ,and a one hour walk at 4.0 mph pace.

SUMMARY:
The purpose of the study is to investigate the acute effect of martial art exercise and aerobic exercise on cognitive performance in college age students. Cognitive performance is a term that encompasses our cognitive processes such as working memory, and executive functioning (decision making); research has found that externally paced (EP) exercise improves cognitive performance and executive functioning (EF). EP activities require decision making skills and higher-level executive functioning. Previous research studies have shown that acute as well as long term aerobic exercise improves cognitive performance Internally paced (IP) exercise requires less attention on task, which may result in less significant improvements in cognitive performance and executive function. However, there is limited research examining the effect that martial art exercise has on these higher-level cognitive functions.Theoretically, the martial art class will improve provide greater stimulation to the higher levels of the brain, causing a greater improvement in the executive function scores when compared to walking. This leads to the question, are externally paced aerobic activities more effective than an acute bout of aerobic exercise in improving executive function in college-aged adults? The investigators hypothesized that martial art training will have a greater impact on executive functioning than aerobic exercise in college-aged adults.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the acute effect of a beginner martial art class and aerobic exercise on cognitive performance in college age students. Cognitive performance is a term that encompasses our cognitive processes such as working memory, and executive functioning (response inhibition); research has found that externally paced (EP) exercise improves cognitive performance and executive functioning (EF). EP activities require decision making skills and higher-level executive functioning. Internally paced (IP) exercise requires less attention on task, which may result in less significant improvements in cognitive performance and executive function. Previous research studies have shown that acute as well as long term aerobic exercise improves cognitive performance. However, there is limited research examining the effect that a martial art class, an external paced exercise, has on these higher-level cognitive functions in college -aged subjects. A study performed by Douris et. al provides a more accurate measure of EP exercise and cognition. Martial arts were used as the complex EP activity. EF in the martial arts group showed greater improvement than the aerobic exercise condition. This was attributed to the complexities of the movement patterns and the associated cortical demands. This study aligns with our current belief that EP activities will have a greater effect than IP activities. The research on the comparison of martial art exercise (externally paced exercise) versus aerobic exercise (internally paced exercise) on executive function is limited to the previous study by the principal investigator utilizing experienced middle-aged martial artists and we presently intend to investigate college aged adults as compared to the previously investigated middle -aged..The current study looks to determine how complex exercise would impact executive functioning. Martial art training requires reactionary movements, quick thinking and decision making, all of which are components of EF. Walking is a relatively simple task that does not require much conscious or cortical control. The investigators plan to have the participants participate in a beginning martial art class and a one hour walk.. Theoretically, the martial art class will improve provide greater stimulation to the higher levels of the brain, causing a greater improvement in the executive function scores when compared to walking. This leads to the question, are externally paced aerobic activities more effective than an acute bout of aerobic exercise in improving executive function in college-aged adults? The proposed research design will be utilizing a randomized cross over repeated measures design. The independent variables are the two one-hour conditions and the dependent variables are the change in Stroop test scores, and stress Visual Analog Scale (VAS) results. In order to test the hypothesis, the investigators will perform a dependent t-test for each dependent variable. An alpha level of p<0.05 will be used for all statistical comparisons. The hypothesis is that an externally paced activity such as martial art exercise will have a greater effect on enhancing executive functioning and will improve stress levels in college aged young adults when compared to an internally paced activity such as walking.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-30 years
* Good overall health
* Exercise at least two days/week

Exclusion Criteria:

* Any cardiopulmonary conditions including asthma within the last 6 months.
* Any major musculoskeletal injuries (i.e. torn ligaments, bone fractures, etc.) over the last 6 months.
* Any other health issues that would interfere with a subject's safety during exercise.
* Any auditory/vestibular impairments.
* Uncorrected visual problems and color blindness.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Executive function | 10 minutes
  For the Stroop tests: the subject will be asked to read words of colors, state the colors of various letters to test processing speed. Subjects will also state the color of the font of a word when the actual word describes a conflicting color. This tests response inhibition, which is a subdivision of executive function. Tower of London which entails a subject is shown the correct organization and is given a specific number of moves to accomplish the task which tests for the problem solving domain of executive function

SECONDARY OUTCOMES:
Stress | 2 minutes
  Visual Analog Scale 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Peter Douris, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: All requests will be reviewed by the principal investigator

REFERENCES:
- [Background] Douris P, Douris C, Balder N, LaCasse M, Rand A, Tarapore F, Zhuchkan A, Handrakis J. Martial Art Training and Cognitive Performance in Middle-Aged Adults. J Hum Kinet. 2015 Oct 14;47:277-83. doi: 10.1515/hukin-2015-0083. eCollection 2015 Sep 29. PMID 26672872
- [Background] Chang YK, Labban JD, Gapin JI, Etnier JL. The effects of acute exercise on cognitive performance: a meta-analysis. Brain Res. 2012 May 9;1453:87-101. doi: 10.1016/j.brainres.2012.02.068. Epub 2012 Mar 4. PMID 22480735
- [Background] Brisswalter J, Collardeau M, Rene A. Effects of acute physical exercise characteristics on cognitive performance. Sports Med. 2002;32(9):555-66. doi: 10.2165/00007256-200232090-00002. PMID 12096929
- [Background] Lee E, Kim Y. Effect of university students' sedentary behavior on stress, anxiety, and depression. Perspect Psychiatr Care. 2019 Apr;55(2):164-169. doi: 10.1111/ppc.12296. Epub 2018 May 24. PMID 29797324
- [Background] Lesage FX, Berjot S, Deschamps F. Clinical stress assessment using a visual analogue scale. Occup Med (Lond). 2012 Dec;62(8):600-5. doi: 10.1093/occmed/kqs140. Epub 2012 Sep 10. PMID 22965867
- [Background] Barella LA, Etnier JL, Chang YK. The immediate and delayed effects of an acute bout of exercise on cognitive performance of healthy older adults. J Aging Phys Act. 2010 Jan;18(1):87-98. doi: 10.1123/japa.18.1.87. PMID 20181996